CLINICAL TRIAL: NCT03631485
Title: An Exploratory Study of Resilience in Parents of Children With Cancer
Brief Title: Exploring the Mental Health of Parents Having Children With Cancer
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 18-371
Record Dates: First submitted 2018-08-07; First posted 2018-08-15 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Resilience of Parents Having Children With Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parents having children with cancer: No intervention.
  Interventions: Other: Exposure_having children with cancer

INTERVENTIONS:
Other: Exposure_having children with cancer — No intervention. The exposure is having children with cancer.

SUMMARY:
Caring for children with cancer is described as life-changing experience and overwhelming stress for parents. Poor quality of life and mental health problems such as depression and anxiety were found in this population. The psychological status of them is still waited to be improved. As a dominant term in positive psychology, resilience is commonly regarded as the ability to move forward or keep normal under adversity. It was proved to be associated with psychological outcomes in adolescents and chronic illness patients, enhanced resilience usually along with improved mental health, while little evidence was available in the parents of children with cancer.

A cross-sectional study will be conducted to explore the level of resilience and psychological outcomes such as quality of life, depression, anxiety and well-being in parents of children with cancer using questionnaires. Such results will be compared with normal population to help evaluate the psychological status of those parents. The relationship between resilience and these psychological outcomes will also be examined. Lower resilience and higher resilience of the parents will be determined by the lowest and highest quartile of The Connor-Davidson Resilience Scale (CD-RISC) scores. Subsequently, a qualitative study will be conducted to explore the experience of those parents with lower resilience and higher resilience.

It is anticipated that risk parents of children with cancer could be identified from the inferior outcomes of resilience and psychological outcomes. Both the results of cross-sectional study and qualitative study will guide the development of interventions designed to enhance resilience and promote positive psychological outcomes among targeted parents of children with cancer under risk.

ELIGIBILITY:
Inclusion Criteria:

* have a child (0-19 years old) with cancer diagnosis. Chinese resident and can read Chinese and speak Mandarin.

Exclusion Criteria:

* have physical impairment or cognitive and learning problems identified from family history of medical records.

attending other researches.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents having children with cancer who are treated at a tertiary hospital in Mainland China between September 2018 and December 2018 will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Resilience measurement by using the Connor-Davidson resilience scale. | A cross-sectional study will be conducted during September 2018 and January 2019. The measurement will be taken once for each participant.
  Resilience of parents having children with cancer will be measured. The total score ranges from 0-100 and higher score reflecting higher level of resilience.

SECONDARY OUTCOMES:
Quality of life measurement by using the Short Form 6D (SF-6D). | A cross-sectional study will be conducted during September 2018 and January 2019. The measurement will be taken once for each participant.
  Quality of life of parents having children with cancer will be measured. The total score ranges from 0.32 for the worst health state to 1 for full health.
Depression measurement by using self-rating depression scale. | A cross-sectional study will be conducted during September 2018 and January 2019. The measurement will be taken once for each participant.
  Depression of parents having children with cancer will be measured. The total score ranges from 20 to 80. Higher total score indicates more serious depression status.
Anxiety measurement by using self-rating anxiety scale. | A cross-sectional study will be conducted during September 2018 and January 2019. The measurement will be taken once for each participant.
  Anxiety of parents having children with cancer will be measured. The total score ranges from 25 to 100 and higher score reflects worse anxiety status.
Stress measurement by using perceived stress scale. | A cross-sectional study will be conducted during September 2018 and January 2019. The measurement will be taken once for each participant.
  Stress of parents having children with cancer will be measured. The total score ranges from 0 to 40. Higher total score suggests more perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Luo Y, Li HCW, Xia W, Cheung AT, Ho LLK, Chung JOK. The Lived Experience of Resilience in Parents of Children With Cancer: A Phenomenological Study. Front Pediatr. 2022 May 30;10:871435. doi: 10.3389/fped.2022.871435. eCollection 2022. PMID 35707743
- [Derived] Luo YH, Li WHC, Cheung AT, Ho LLK, Xia W, He XL, Zhang JP, Chung JOK. Relationships between resilience and quality of life in parents of children with cancer. J Health Psychol. 2022 Apr;27(5):1048-1056. doi: 10.1177/1359105321990806. Epub 2021 Jan 31. PMID 33522296